CLINICAL TRIAL: NCT05677607
Title: Feedback Loop Between Intracranial Atherosclerosis and Cerebral Small Vessel Disease
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jinhao Lyu, Attending physician, Chinese PLA General Hospital
Other Study IDs: 301Brainmax
Record Dates: First submitted 2022-12-19; First posted 2023-01-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: ICAS - Intracranial Atherosclerosis; Cerebral Small Vessel Diseases
Keywords: Intracranial atherosclerosis; Cerebral small vessel disease; Feedback mechanism; Multimodal MRI
MeSH Terms: conditions — Intracranial Arteriosclerosis; Cerebral Small Vessel Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intracranial atherosclerosis and small vessel disease: Patients diagnosed with intracranial large artery atherosclerosis and cerebral small vessel disease based on imaging screening.
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — Imaging diagnostics mainly based on Magnetic resonance imaging.

SUMMARY:
The present study aims at verifying the mutual effects between intracranial large artery atherosclerosis and cerebral small vessel disease on disease progression and prognosis by magnetic resonance imaging, and providing biomarkers for the early prevention and treatment of cerebrovascular disease.

DETAILED DESCRIPTION:
Cerebrovascular disease is the most common cause of death worldwide. There is a close link in structure and function between the intracranial large arteries and cerebral small vessels. Moreover, growing evidences have demonstrated that large artery atherosclerosis often coexists with small vessel disease, which may deteriorate the clinical outcomes of stroke and dementia. The mutual feedback mechanism between them is not fully understood. The present study focuses on the mechanism of mutual feedback between large artery atherosclerosis and cerebral small vessel disease by using magnetic resonance imaging. The study may provide biomarkers for the early prevention and treatment of cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* At least one intracranial artery ≥ 50% atherosclerotic stenosis
* Modified Rankin Scale < 2
* Mini-mental State Examination > 24

Exclusion Criteria:

* Concurrent ipsilateral extracranial artery ≥ 50% stenosis
* Pregnant women
* Contraindications to magnetic resonance examination (patients with pacemakers, nerve stimulators, artificial metal heart valves and other metal foreign bodies)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with at least on intracranial artery ≥ 50% atherosclerotic stenosis.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression in total cerebral small vessel disease burden | 1-3 YEARS
  Total cerebral small vessel disease burden is assessed according to a sum of scores of white matter hyperintensity, cerebral microbleeds, lacunes and enlarged perivasular spaces on magnetic resonance imaging sequences.
Frequency of stroke recurrence | 1-3 YEARS
  The percentage of symptomatic participants who suffer from stroke recurrence after enrollment in the territory of the targeted stenotic vessel.

SECONDARY OUTCOMES:
Frequency of stroke of asymptomatic participants | 1-3 YEARS
  The percentage of asymptomatic participants who suffer from stroke after enrollment in the territory of the targeted stenotic vessel.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhao Lyu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No